CLINICAL TRIAL: NCT03940729
Title: People Who Inject Drugs; Longitudinal Staphylococcus Aureus Colonization Pattern and the Impact on Infection Frequency by Regular Showers With Chlorhexidine
Brief Title: PWID; Longitudinal S Aureus Colonization Pattern and the Impact on Infection Frequency by Regular Showers With Chlorhexidine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Intravenous Drug Abuse, S Aureus Colonization
Keywords: PWID; S aureus; colonization; infection; chlorhexidine
MeSH Terms: conditions — Substance Abuse, Intravenous; Staphylococcal Infections; Infections | interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PWID colonized with S aureus (Other): Repeated chlorhexidin showers for PWID colonized with S aureus
  Interventions: Drug: Chlorhexidine Topical

INTERVENTIONS:
Drug: Chlorhexidine Topical — In the Malmö needle exchange program, people who inject drugs (PWID) are repeatedly screened for S aureus colonization during one year. Those colonized will repeatedly shower with chlorhexidine during the following year. The infection frequency will be compared between the two periods.

SUMMARY:
People who inject drugs (PWID) have increased risk of Staphylococcus aureus (S. aureus) colonization, skin and soft tissue infections (SSTI), and systemic infections like septicaemia and endocarditis. International research and data from Malmö needle exchange program (NEP) show a 60 - 70% lifetime SSTI prevalence. Longitudinal colonization pattern of S. aureus and its association with infection frequency among PWID is unknown. Cultures from the anterior nares, throat and perineum are used to indirectly assess S. aureus skin colonization. In PWID 28 - 45% are colonized in the nares, which increases risk of infections. Clinical significance of extra-nasal colonization, and persistent/intermittent colonization is uncertain.

The S. aureus genome can be characterized by whole genome sequencing (WGS). Certain types are associated with abscesses and systemic infections. The infection pattern among PWID is unknown.

S. aureus skin colonization level is decreased by chlorhexidine body wash and nasal mupirocin used as surgical prophylaxis and treatment of furunculosis. To our knowledge, disinfection effect on infections in PWID is not studied. However, the clinical impression is that severe infections have somewhat diminished since the NEP started distributing skin disinfectant tissues.

RESEARCH QUESTIONS

1. Can repeated skin wash with chlorhexidine decrease infection frequency among PWID?
2. Is the longitudinal S. aureus colonization pattern associated with infection prevalence among PWID?
3. Can the risk of S. aureus-infections be predicted by quantification of bacterial level in anterior nares, throat, perineum or skin lesions/eczema?
4. Can different types of S. aureus be identified, that are associated with colonization or infection among PWID (by WGS)?

METHODS AND TIME PHRAME Malmö NEP was established in 1986, and several studies assessing HIV, hepatitis and sociological questions have been conducted in this setting. In December 2016 continuous inclusion of 100 PWID for the actual study started at Malmö NEP. The study period is estimated to two years, with scientific papers expected for publication.

During the first year of the study, mapping of S. aureus colonization pattern among all study participants is conducted by repeated sampling, clinical evaluation of eczemas, and interviews regarding infections. Every third month samples are collected from nares, throat, perineum and skin lesions. Semi quantification of S. aureus takes place at the microbiological research laboratory at Lund University. BBL CHROMagar Staph aureus-plates are used and incubated in 35oC air for 48h. S. aureus-colonies are identified and quantified manually by pink colour change and Pastorex. MALDI-TOF will be used in unclear cases. Disk-diffusion will be used for resistance determination. Bacterial isolates will be frozen to -70oC for later WGS.

Intervention with chlorhexidine wash starts one year after inclusion for each study subject, and will continue for one additional year. Study participants with S aureus colonization will undergo regular showers with chlorhexidine (intervention group) at the needle exchange. In order to avoid bacterial resistance, muporicin will not be used. During the intervention, cultures, interviews and clinical evaluation will continue.

ELIGIBILITY:
Inclusion Criteria: Participants in a needle exchange program who are willing to undergo study procedures -

Exclusion Criteria: No

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Infection frequency | Two years
  Infections are regularly evaluated through interviews and Medical record reviews

SECONDARY OUTCOMES:
Hospital admittance | Two years
  Evaluated through medical records
Antibiotic prescription | Two years
  Evaluated through medical records
Death | Two years
  Evaluated through medical records

CONTACTS AND LOCATIONS:
Overall Officials: Maria Josephson, MD, Study Director — VO Infektionssjukdomar SUS

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers